CLINICAL TRIAL: NCT03647046
Title: Custom Anterior Surfacing of Scleral Lens for Vision Quality Improvement in Patients With Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Ovitz Corporation (Industry); Boston Sight (Other)
Responsible Party: Principal Investigator, Tara Vaz, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 72749
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-12

CONDITIONS: Keratoconus
Keywords: Keratoconus, scleral lens
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Customized Scleral Lens (Experimental): A customized scleral lens will be compared with a non-customized scleral lens in subjects with Keratoconus through vision tests.
  Interventions: Device: Customized Scleral Lens

INTERVENTIONS:
Device: Customized Scleral Lens — A wavefront customized scleral lens will be made for each subject and tested against a non-customized lens.

SUMMARY:
The goal of the study is to examine the effects of custom front-surface wavefront correction on visual performance, and on neutralization of higher order aberrations, in patients wearing a scleral lens device. The investigators will study patients with keratoconus, the most common type of corneal ectasia, who have already been fitted with the BostonSight BSS (Boston Sight Scleral) for improved visual function.

DETAILED DESCRIPTION:
This study will be a single center, double-masked collection of data taking place at the Flaum Eye Institute. Informed consent will be obtained from all subjects after a thorough explanation of the nature and possible risks of the study. Flaum Eye Institute electronic health records of existing patients will first be screened by an optometrist or ophthalmologist to verify that they do not fall under the exclusion criteria. Some study communication regarding scheduling will be done over the phone or email. The screening will be similar to a standard eye exam (without eye dilation) and will include a slit lamp examination as well as visual acuity and basic vision evaluation.

The study eye will be chosen based on inclusion criteria; if both eyes qualify, the eye with worse best corrected acuity will be chosen. A new lens will be manufactured for the subject after the screening visit and will be given to the subject during the following study visit. This is done to ensure fully neutralized spherical refractive effort and positional stability. If screening evaluation reveals that the current lens does not fully neutralize spherical refractive error or that the current lens is not positionally stable, a baseline lens will be manufactured that corrects this. The subject will be allowed to keep the old lens if he or she so chooses.

At the second visit, the patient's vision and fit will be evaluated with the optimized baseline BSS lens. Visual acuity and device fit will be evaluated and recorded. If the BSS device fit is still not optimized, then a new device will be made , and the second visit evaluation will be rescheduled. Once the baseline lens design is determined to be satisfactory, the patient will have their wavefront aberration measured with a wavefront sensor. Investigators will dilate the pupil pharmacologically with phenylephrine (2.5%) and tropicamide (1%) and take wavefront measurements of the optical aberrations of the subject's eye wearing the baseline lens using a portable, non-invasive wavefront analyzer designed to measure highly aberrated eyes (Ovitz, P10/EyeProfiler). The investigators will then design and manufacture a study lens that is identical in design to the baseline BostonSight BSS lens except for a custom front surface designed to neutralize the optical aberrations measured with the wavefront analyzer. This HOA-optimized lens will be created prior to the third visit.

At the third visit the patient's vision and fit will be evaluated with the new HOA-optimized lens. A designated study team member will measure visual acuity and over-refraction of the patient. If an adjustment is needed for the lens, then a new device will be made, and the third visit evaluation will be rescheduled.

Once well-fitting baseline and HOA-optimized test lenses are established, both lenses will be remade and presented to the evaluator designated study team member in charge of evaluation and subject together in a masked fashion. During a fourth visit, the patient's vision will be extensively evaluated using standard non-invasive optometric measurements with each of the two lenses. First the patient will undergo a basic evaluation with each lens to ensure that the fit is correct. The patient will then undergo basic visual acuity; high and low contrast visual acuity, contrast sensitivity, and subjective vision scoring with each lens. The subject's wavefront aberration will also be measured again with each lens.

ELIGIBILITY:
A person will be included in the study if he/she:

* Is 18 years or older and has full legal capacity to volunteer.
* Has been diagnosed with Keratoconus;
* Has no other active ocular disease;
* Is currently wearing the BostonSight BSS in at least one eye ;
* Has non-spherical BostonSight BSS haptic design in the study eye;
* Has 20/400 or better best corrected visual acuity with pinhole 20/60 or better in the study eye;
* Is not pregnant or nursing;
* Has voluntarily agreed to participate in the study by signing the statement of informed consent;

A person will be excluded from the study if he/she:

* Is under the age of 18;
* Has best corrected visual acuity outside 20/400;
* Pregnant or nursing at the time of enrollment in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Flaum Eye Institute, University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Customized Scleral Lens
Started | 12
Completed | 8
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Customized Scleral Lens
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 40.9 [20 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Keratoconus [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal Vision
Description: Vision will be tested using the Basic Snellen Visual Acuity test and normal vision will be defined as 20/20.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Customized Scleral Lens
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Customized Scleral Lens
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT03647046/Prot_SAP_001.pdf
  • Informed Consent Form (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03647046/ICF_002.pdf